CLINICAL TRIAL: NCT00514241
Title: A Clinical Study to Evaluate the Use of Gravitational Platelet Separation System on Leg Wound Healing in Coronary Bypass Surgery
Brief Title: Evaluate Use of Gravitational Platelet Separation System on Leg Wound Healing in Coronary Bypass Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JA-250-N
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Coronary Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- A (Experimental): The arm utilizes the GPS™ II Platelet Concentrate Separation Kit.
  Interventions: Device: The GPS™ II Platelet Concentrate Separation Kit
- B (No Intervention): This arm utilizes standard leg wound closure procedures.

INTERVENTIONS:
Device: The GPS™ II Platelet Concentrate Separation Kit — The GPS™ II Platelet Concentrate Separation Kit system is designed to be used for the safe and rapid preparation of autologous platelet-rich-plasma (PRP) from a small sample of blood at the patient's point of care. The PRP can be mixed with autograft and allograft bone prior to application to an orthopedic surgical site as deemed necessary by the clinical use requirements.
  Arms: A

SUMMARY:
The aim of platelet rich plasma (PRP) application is to accelerate the healing cascade via application of elevated cytokine concentrations released during platelet degranulation.

This is a prospective randomized study of the effect of autologous platelet concentrate application during surgical closure following a vein harvest during coronary bypass surgery. This prophylactic measure will be compared to standard surgical closure techniques with the primary outcome being the incidence of leg wound infection.

DETAILED DESCRIPTION:
Postoperative wound disturbances, particularly surgical site infection of the chest and leg incision site following cardiac surgery are associated with increased morbidity, mortality, and costs. A recent dissertation from the National hospital in Norway showed a 20% infection rate in wounds after bypass surgery, this is probably representable nation wide. Prophylactic interventions that reduce postoperative wound disturbances and infection would have inherent value in cardiothoracic surgery. Ideally, a specific intervention would demonstrate improved patient outcomes while reducing the output of hospital resources.

The aim of platelet rich plasma (PRP) application is to accelerate the healing cascade via application of elevated cytokine concentrations released during platelet degranulation. It is hypothesized that the elevated cytokine levels will elucidate an accelerated healing response of the affected tissue. PPP application has also been advocated as a tissue sealant for topical hemostasis.

This is a prospective randomized study of the effect of autologous platelet concentrate application during surgical closure following a vein harvest during coronary bypass surgery. This prophylactic measure will be compared to standard surgical closure techniques with the primary outcome being the incidence of leg wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a cardiothoracic procedure requiring a leg vein harvest
* Patient signature of informed consent form

Exclusion Criteria:

* Pregnancy
* < 18 years of age
* History of amenia (hemoglobin < 11.0)
* History of bleeding disorder
* Un-cooperative patient or patient with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations
* Hypothyroidism
* History of any blood disorder
* Patient with an active infection
* Patients taking Cox II inhibitors.
* Heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Presence/absence of leg wound infection, General wound healing - picture evaluation | 6 weeks

SECONDARY OUTCOMES:
ASEPSIS Score, Length of hospital stay, Reoperation rate for bleeding and infection control | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fredrik Stray, B. Sc, MBA, Principal Investigator — Biomet Norge A.S.
Locations (1):
- Feiringklinikken AS, Feiring, Norway

IPD SHARING:
Plan to Share IPD: No